CLINICAL TRIAL: NCT01100515
Title: Phase 3 Study of Hyperbaric Oxygen Therapy in Non-Comatose Patients With Acute Domestic Carbon Monoxide Poisoning
Brief Title: Hyperbaric Oxygen Therapy for Acute Domestic Carbon Monoxide (CO) Poisoning
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: this study was suspended for futility
Sponsor: University of Versailles (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Christophe Misse, DRRC Assistance Publique Hôpitaux de Paris
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CO89
Record Dates: First submitted 2010-04-05; First posted 2010-04-09 (Estimated); Last update posted 2010-04-09 (Estimated); Status verified 2010-04

CONDITIONS: Carbon Monoxide Poisoning
Keywords: intoxication; carbon monoxide; adults; domestic accident; acute domestic carbon monoxide poisoning
MeSH Terms: conditions — Carbon Monoxide Poisoning | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental arm (Experimental): Hyperbaric oxygen therapy at 2 absolute atmosphere (1-hour plateau) followed by 4 hours of normobaric oxygen therapy
  Interventions: Other: Hyperbaric oxygen therapy
- Control (Active Comparator): 6 hours course of normobaric oxygen therapy via a face full mask
  Interventions: Other: normobaric oxygen therapy

INTERVENTIONS:
Other: normobaric oxygen therapy — oxygen therapy was delivered via a full face mask at high flow to achieve 100% of inspired oxygen fraction
  Arms: Control
Other: Hyperbaric oxygen therapy — Hyperbaric oxygen therapy was delivered in a hyperbaric chamber, pressurized at 2 absolute atmosphere (1 hour plateau) and the patient breathed high oxygen concentration via a full face mask followed by 4 hours of normobaric oxygen therapy
  Arms: Experimental arm

SUMMARY:
Carbon monoxide poisoning still places a burden on the healthcare system worldwide. While oxygen therapy is the cornerstone treatment, the role and practical modalities of hyperbaric oxygen therapy (HBO) remain controversial. This study aimed at comparing one session of HBO at 2 absolute atmosphere followed by 4 hours of normobaric oxygen therapy to 6 hours of normobaric oxygen therapy in adult victims of acute domestic carbon monoxide poisoning and without coma.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 15 years of age
* admitted for domestic CO poisoning within 12 hours after the end of CO exposure.
* had transient loss of consciousness (syncope, malaise)
* carboxyhemoglobin level at presentation >10% or 5%, in smokers and non-smokers, respectively.

Exclusion Criteria:

* poisoning by more than one compound (e.g., CO plus a drug or CO plus other toxic gases such as those found in fire smoke
* suicide attempt
* pregnancy
* coma
* contraindications to HBO (circulatory collapse or pneumothorax)
* technical obstacles to HBO
* non domestic CO poisoning
* difficulty in determining whether the patient experienced initial loss of consciousness or initial coma
* consent refusal.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 1989-10; Primary Completion 2000-01 (Actual); Study Completion 2000-02 (Actual)

PRIMARY OUTCOMES:
full recovery | at one month
  Full recovery was defined as an absence of symptoms reported on the self-assessment questionnaire with a normal physical exam (including normal neuropsychological functions).

SECONDARY OUTCOMES:
persistent neurological sequels | at one month
  Neurological sequels were considered persistent (PNS) if they were present both at hospital discharge and at one-month evaluation, regardless of the type of manifestation
delayed neurological sequels | at one month
  Delayed neurological sequelae (DNS) were any neurological manifestations that appeared between hospital discharge and one-month evaluation, regardless of their severity. Patients with DNS were those considered fully recovered at hospital discharge but with neurological manifestations at one-month evaluation
variations in carboxyhemoglobin levels | at 12 hours from randomization
  the difference in serum carboxyhemoglobin levels between baseline values and values recorded immeadiately after study treatment completion
serious adverse events | at one month
  any complications of hyperbaric oxygen therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Raymond Poincaré Hospital, Garches, France